CLINICAL TRIAL: NCT02026947
Title: Sodium Benzoate for Treatment of Attenuated/Transient Psychosis. A Randomized Placebo-controlled Trial.
Acronym: AttenPsyc
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We did not commence the trial because there were no patients who could fulfill the inclusion criteria.
Sponsor: Niuvanniemi Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jari Tiihonen, Professor, Niuvanniemi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3418363; 2013-000458-23 (EudraCT Number)
Record Dates: First submitted 2013-12-27; First posted 2014-01-03 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Attenuated or Transient Psychosis
MeSH Terms: interventions — Sodium Benzoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In both arms, one capsule at the morning for the first week. One capsule at the morning and one at the evening for the weeks 2-12.
  Interventions: Drug: Placebo
- Sodium benzoate (Experimental): 0.5 g/day during the first week, 1.0 g/day for the next 11 weeks. One capsule at the morning for the first week. One capsule at the morning and one at the evening for 2-12 weeks.
  Interventions: Drug: Sodium Benzoate; Drug: Placebo

INTERVENTIONS:
Drug: Sodium Benzoate — 0.5 g/day during the first week, 1.0 g/day for the next 11 weeks. One capsule at the morning for the first week. One capsule at the morning and one at the evening for 2-12 weeks.
  Arms: Sodium benzoate
Drug: Placebo

SUMMARY:
The aim of this study is to investigate whether sodium benzoate is superior to placebo in decreasing symptoms among patients with attenuated/transient psychosis. A total of 140 patients will be randomized in 1:1 ratio to receive sodium benzoate 1 g/day or placebo for 12 weeks. Concerning statistical power, the number of patients is sufficient to obtain statistical significance for a clinically meaningful effect size of 0.40 (Cohen's d). The primary outcome measure is change in PANSS sum score of delusions, hallucinations, suspiciousness and conceptual disorganization (the PANSS items that are inclusion criteria) at week 12. Change in CGI score at week 12 is the other primary outcome measure. The secondary outcome measures are change in PANSS total score at week 12, CGI score at week 24, and GAF at weeks 12 and 24.

DETAILED DESCRIPTION:
Early treatment of psychotic disorders results in better outcome, and several small randomized controlled trials (RCTs) have indicated that pharmacological treatment of prodromal patients with subthreshold psychosis might prevent transition to psychotic disorders. Use of risperidone had statistically significant effect at 6 months, but not at 12 months, and olanzapine has shown only a beneficial trend. The use of antipsychotics for the prevention of psychosis is controversial due their adverse effects and, therefore, use of better-tolerated agents such as natural compounds like benzoid acid or omega fatty acids might be a promising approach.

Glutamatergic hypothesis has gained increasing support explaining symptoms of schizophrenia, and hypofunction of N-methyl-D-aspartate (NMDA) receptor is considered nowadays a major factor in the pathophysiology of the disease. Several NMDA-enhancing agents such as glycine, D-alanine, D-serine, sarcosine and bitopertin have shown beneficial effect as add-on treatments to antipsychotics. D-amino acid oxidase (DAAO) metabolizes D-alanine and D-serine, which are co-agonists of NMDA-receptor, and, therefore, decreasing DAAO activity results into enhancement of NMDA-receptor function. Recently, a randomized controlled trial in 52 patients with chronic schizophrenia was well tolerated and showed a robust beneficial effect of DAAO inhibitor sodium benzoate (1 g/d) as compared with placebo (effect size 1.76 for PANSS total scores; Tsai et al. 2012).

The aim of this study is to investigate whether sodium benzoate is superior to placebo in decreasing symptoms among patients with attenuated/transient psychosis. A total of 140 patients will be randomized in 1:1 ratio to receive sodium benzoate 1 g/day or placebo for 12 weeks. Concerning statistical power, the number of patients is sufficient to obtain statistical significance for a clinically meaningful effect size of 0.40 (Cohen's d). The primary outcome measure is change in PANSS sum score of delusions, hallucinations, suspiciousness and conceptual disorganization (the PANSS items that are inclusion criteria) at week 12. Change in CGI score at week 12 is the other primary outcome measure. The secondary outcome measures are change in PANSS total score at week 12, CGI score at week 24, and GAF at weeks 12 and 24.

An interim analysis will be done after obtaining results from the first 40 patients. If the effect size (Cohen's d) for primary outcome measures is less than 0.30, the study will be stopped prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Age is from 15 to 30 years
* Meet at least 1 criteria for either of following groups:

Group a. Attenuated Psychotic Symptoms: Symptom scores of 3 on the PANSS delusions scale, 2-3 on the PANSS hallucinations scale, 3-4 on PANSS suspiciousness, or 3-4 on PANSS conceptual disorganization scale (frequency of symptoms ≥ 2 times/wk for a period of at least 1 week and not longer than 5 years, to have occurred within the last year)

Group b. Transient Psychosis: Symptoms scores of ≥ 4 on PANSS hallucinations scale, ≥ 4 on PANSS delusions scale, or ≥ 5 on PANSS conceptual disorganization scale (symptoms not sustained beyond a week and resolved without antipsychotic medication within the last year)

Exclusion Criteria:

* a history of a previous psychotic disorder or manic episode (both treated or untreated);
* substance-induced psychotic disorder;
* acute suicidal or aggressive behavior;
* a current DSM-IV diagnosis of substance dependence (except cannabis dependence);
* neurological disorders (e.g., epilepsy);
* IQ of less than 70 (no diagnosis of mental retardation as verified by school performance);
* previous treatment with an antipsychotic or mood-stabilizing agent (>1 week);
* pregnancy or inadequate pregnancy prevention among sexually active females,
* history of allergy or severe adverse events for sodium benzoate;
* laboratory values more than 10% outside the normal range for transaminases, thyroid hormones, or C-reactive protein; and
* another severe intercurrent illness that may have put the person at risk or influenced the results of the trial or affected their ability to take part in the trial. Use of benzodiazepine-derivatives is allowed during the trial.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change in PANSS sum score of delusions, hallucinations, suspiciousness, and conceptual disorganization | baseline - week 12
  change in PANSS sum score of delusions, hallucinations, suspiciousness and conceptual disorganization (the PANSS items that are inclusion criteria)
change in Clinical Global Improvement Scale (CGIS) | baseline - week 12

SECONDARY OUTCOMES:
change in Clinical Global Improvement (CGI) | baseline - week 24
change in Positive and Negative Syndrome Scale (PANSS), Total score | baseline - week 12
change in Global Assessment of Functioning (GAF) | baseline - weeks 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Jari Tiihonen, MD, PhD, Principal Investigator — Niuvanniemi Hospital
Locations (2):
- Finland (2):
  - HUS Health Care District, Helsinki
  - Varsinais-Suomi and Satakunta Health Care District, Turku